CLINICAL TRIAL: NCT04775836
Title: A Platform for Linking and Assessing To Facilitate Outcomes and Research Methods in CerebroVascular Diseases Using Electronic Health Records (PLATFORM-CVD)
Brief Title: An EHR-based Platform To Facilitate Outcomes and Research Methods in Cerebrovascular Diseases
Acronym: PLATFORM-CVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Dalian Jiuzhou Century Hospital (Unknown); Dengzhou Central Hospital (Unknown); Guangxi Ruikang Hospital (Other); Guangdong Second Provincial General Hospital (Other); Handan Central Hospital (Other); Xunxian People's Hospital (Unknown); Kaifeng Central Hospital (Other); Laoling People's Hospital (Unknown); New Area People's Hospital of Luoyang (Unknown); Chinese Traditional Medicine Hospital of Meishan (Unknown); Mengjin People's Hospital (Unknown); Nanyang Central Hospital (Other); Hexigten Banner Mongolian Traditional Chinese Medicine Hospital (Unknown); Inner Mongolian Hospital of Traditional Chinese Medicine (Unknown); The Affiliated Hospital of Qingdao University (Other); Renqiu Kangjixintu Hospital (Unknown); Shenzhen Second People's Hospital (Other); Wuhan No.1 Hospital (Other); Xingtai City Ninth Hospital (Unknown); Yilong People's Hospital (Unknown); Yongcheng City Central Hospital (Unknown); Chongqing Donghua Hospital (Unknown); The Second Affiliated Hospital of Luohe Medical College (Unknown)
Responsible Party: Principal Investigator, Yongjun Wang, MD, Professor, Ministry of Science and Technology of the People´s Republic of China
Other Study IDs: 2017YFC1310901
Record Dates: First submitted 2021-02-05; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Cerebrovascular Diseases; Cerebral Infarction; Cerebral Hemorrhage; Transient Ischemic Attack; Subarachnoid Hemorrhage
Keywords: Healthcare Quality; Electronic Health Records; Cerebrovascular Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Cerebral Infarction; Cerebral Hemorrhage; Ischemic Attack, Transient; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this protocol, the investigators present methods and preliminary results from the PLATFORM-CVD Study, an EHR-based multicenter cohort. This study will focus on assessing the distribution of major cerebrovascular diseases, determining the risk factors associated with disease incidence and worse in-hospital outcomes, as well as describing the quality of care. Data from this cohort will be used to develop suitable prediction models for cerebrovascular diseases using real-world data and to understand how outcomes for cerebrovascular diseases would change with quality improvement interventions.

DETAILED DESCRIPTION:
Adherence to healthcare quality measures is needed to reduce the burden of cerebrovascular disease and improve clinical outcomes. Electronic health records (EHRs) can facilitate the standardization of care provision and the improvement of disease prediction and prevention. Although the EHRs in clinical settings are increasingly prevalent in China, they are rarely used for healthcare research. the investigators aimed to conduct an EHR-based registry study to improve the healthcare and outcomes for cerebrovascular diseases.

Twenty-four hospitals were enrolled in the PLATFORM-CVD Study in January 2018. Data collection began on February 1st, 2019. Historical data from January 2017 are abstracted first and prospective data are continuously reported until May 20th, 2020. Data were abstracted from the medical records, including hospital information system, laboratory information management system, and picture archiving and communication systems by an extract-transform-load tool. The EHR system included diagnostic information for cerebral infarctions (I63), nontraumatic intracerebral hemorrhages (I61), nontraumatic subarachnoid hemorrhages (I60), transient cerebral ischemic attacks and related syndromes (G45), intracranial and intraspinal phlebitis and thrombophlebitis (G08), vascular dementia (F01), and other aneurysms (I72). The quality of stroke care was assessed by 21 evidence-based performance measures. In-hospital outcomes were calculated including mortality, length of stay, and costs.

The PLATFORM-CVD Study leverages EHRs to better understand incident cerebrovascular diseases in China. Data from this cohort will serve as a unique platform for quality assessment and improvement for acute treatment and secondary prevention of cerebrovascular diseases, as well as in-hospital outcome risk predictions and health economic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the registry if they were hospitalized with a primary diagnose of：
* cerebral infarction (I63)
* nontraumatic intracerebral hemorrhage (I61)
* nontraumatic subarachnoid hemorrhage (I60)
* transient cerebral ischemic attack and related syndromes (G45)
* intracranial and intraspinal phlebitis and thrombophlebitis (G08)
* vascular dementia (F01)
* other aneurysms (I72)

Exclusion Criteria:

* Patients diagnosed with other diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty-five hospitals were enrolled in the PLATFORM-CVD Study between January 1st, 2017 and May 20th, 2020. Hospitals were included if they: 1) had neurological wards; 2) were secondary or tertiary hospitals; 3) could admit at least 20 cerebrovascular disease patients every month.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | From date of hospitalization until the date of discharge, assessed up to 90 days
  Patients who died during hospitalization due to cerebrovascular diseases
Length of stay at hospital | From date of hospitalization until the date of discharge, assessed up to 90 days
  The total days for a patients with cerebrovascular diseases at hospitalization
Costs | From date of hospitalization until the date of discharge, assessed up to 90 days
  The total costs for a patients with cerebrovascular diseases at hospitalization

SECONDARY OUTCOMES:
Rate of antiplatelet medication use | From date of hospitalization until the date of discharge, assessed up to 90 days
  Rate of antiplatelet therapy during hospitalization
Rate of dual antiplatelet medication use for non-disabling IS and TIA events | From date of hospitalization until the date of discharge, assessed up to 90 days
  Rate of aspirin and clopidogrel therapy for ischemic cerebrovascular diseases (IS or TIA) during hospitalization
Rate of DVT prophylaxis ≤ 48 hours | 48 hours within hospitalization
  Patients at risk for DVT (non-ambulatory) who received DVT prophylaxis by end of hospital 48 hours, including pneumatic compression, warfarin sodium, and novel oral anticoagulant
Cerebrovascular assessment ≤ seven days | 7 days within hospitalization
  Cerebrovascular assessment (TCD, IVUS, brain CT or MR scan) within seven days of hospitalization
Statin therapy for LDL ≥100 mg/dL during hospitalization | From date of hospitalization until the date of discharge, assessed up to 90 days
  Lipid lowering agent prescribed during hospitalization if LDL ≥ 100 mg/dL, if patient treated with lipid lowering agent prior to admission, or LDL not documented
Rate of anticoagulation medication use for atrial fibrillation during hospitalization | From date of hospitalization until the date of discharge, assessed up to 90 days
  Anticoagulation prescribed during hospitalization in patients with documented atrial fibrillation
Rate of antithrombotic medication prescribtion at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Antithrombotic therapy prescribed at discharge, including antiplatelet or anticoagulant therapy
Rate of antihypertensive medication prescribtion for patients with hypertension at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Antihypertension medication prescribed at discharge for patients with history of hypertension disease or hypertension disease documented during the hospitalization
Rate of statin prescribtion for low-density lipoprotein≥100 mg/dL at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Lipid lowering agent prescribed at discharge if LDL ≥ 100 mg/dL, if patient treated with lipid lowering agent prior to admission, or LDL not documented
Rate of hypoglycaemia medication prescribtion for diabetes mellitus at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Hypoglycemic medication prescribed at discharge for patients with history of diabetes mellitus or diabetes mellitus documented during the hospitalization
Rate of anticoagulation medication prescribtion for atrial fibrillation at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Anticoagulation prescribed at discharge in patients with documented atrial fibrillation
Rate of thrombolytic therapy | From date of hospitalization until the date of discharge, assessed up to 90 days
  Intravenous r-tPA in IS patients
Rate of thrombectomy therapy | From date of hospitalization until the date of discharge, assessed up to 90 days
  Thrombectomy therapy for IS patients
Rate of DVT prophylaxis ≤ 48 hours for ICH | 48 hours within hospitalization
  Patients with ICH at risk for DVT (non-ambulatory) who received DVT prophylaxis by end of hospital 48 hours, including pneumatic compression.
Rate of antihypertensive medicine use for ICH patients with hypertension at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Antihypertension medication prescribed at discharge for ICH patients with history of hypertension disease or hypertension disease documented during the hospitalization
Rate of hypoglycemia medication use for ICH patients with diabetes mellitus at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Hypoglycemic medication prescribed at discharge for ICH patients with history of diabetes mellitus or diabetes mellitus documented during the hospitalization
Rate of neurosurgery for ICH patients | From date of hospitalization until the date of discharge, assessed up to 90 days
  Neurosurgery of ICH include removal of hematoma by craniotomy, aspiration of hematoma by drilling, decompressive craniectomy, ventriculocentesis and drainage, other removal of intracranial hematoma
Rate of DVT prophylaxis ≤ 48 hours for SAH | 48 hours within hospitalization
  Patients with SAH at risk for DVT (non-ambulatory) who received DVT prophylaxis by end of hospital 48 hours, including pneumatic compression
Rate of antihypertensive medicine use for SAH patients with hypertension at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Antihypertension medication prescribed at discharge for SAN patients with history of hypertension disease or hypertension disease documented during the hospitalization
Rate of hypoglycemia medication use for SAH patients with diabetes mellitus at discharge | From date of hospitalization until the date of discharge, assessed up to 90 days
  Hypoglycemic medication prescribed at discharge for SAH patients with history of diabetes mellitus or diabetes mellitus documented during the hospitalization
Rate of neurosurgery for SAH patients | From date of hospitalization until the date of discharge, assessed up to 90 days
  Neurosurgery of SAH include aneurysm clipping, endovascular embolization of aneurysm, extraventricular shunt

CONTACTS AND LOCATIONS:
Overall Officials: Zi-Xiao Li, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share the data dictionary of the study. The data could be applied by the PI's email. Applicant should make an SAP first. The PI will check the SAP and appoint a statistician for the analysis.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available when the data collection finished.